CLINICAL TRIAL: NCT06337331
Title: A Phase II Trial of Venetoclax-Enhanced Reduced Intensity HLA-Mismatched Allogeneic Transplant for Ultra-High-Risk Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Brief Title: Adding Venetoclax to the High-dose Chemotherapy Regimen Prior to Mismatche Allogeneic Stem Cell Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to accommodate FDA recommendations for protocol revisions
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 1401
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — venetoclax; Decitabine; fludarabine; Busulfan; Whole-Body Irradiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- High-dose Chemotherapy + Mismatched Allogeneic Stem Cell Transplant (Experimental)
  Interventions: Drug: Venetoclax; Drug: Decitabine; Drug: Fludarabine; Drug: Busulfan; Radiation: Total Body Irradiation

INTERVENTIONS:
Drug: Venetoclax — 400mg/day PO Days -8 to -2
Drug: Decitabine — 20mg/m2/day IV Days -7 to -3
Drug: Fludarabine — 30mg/m2/day IV Days -7 to -3
Drug: Busulfan — 3.2mg/kg/day IV Days -5 to -4
Radiation: Total Body Irradiation — 200cGy Day -2

SUMMARY:
Patients eligible for a mismatch allogeneic stem cell transplant will receive Venetoclax daily for 7 days prior to transplant in addition to the following chemotherapy regimen: Decitabine daily for 5 days, Fludarabine daily for 5 days, and Busulfan daily for 2 days followed by 1 day of total body irradiation. Stem cell transplant will occur thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Availability of a 4/8 - 6/8 HLA-matched related donor or a 7/8 HLA-matched unrelated donor
* Receiving first allogeneic transplant
* KPS >/= 70%
* MDS associated with TP53 mutation AND R-IPSS high or very high risk at diagnosis OR
* AML with adverse risk cytogenetics or molecular abnormalities according to the 2017 ELN risk stratification OR pre-transplant MRD by either flow cytometry, cytogenetics or FISH
* Less than 5% myeloblasts in the marrow pre-transplant

Exclusion Criteria:

* Poor cardiac function defined as LVEF <45%
* Poor pulmonary function defined as FEV1, FVC, or DLCO <50% predicted
* Poor liver function defined as bilirubin >/=2.5mg/dL, AST/ALT >3xULN
* Poor renal function defined as creatinine >/=2.0mg/dL or CrCl <40mL/min
* Ongoing or active systemic infection, active Hepatitis B or C virus infection, or known HIV positivity
* Patient requiring treatment with a moderate or strong inhibitor or inducer of CYP3A4 or a P-gp inhibitor within 7 days prior to starting preparative chemotherapy through Day +4 post-transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of relapse/progression by conducting blood and bone marrow biopsy evaluations at one-year post-transplant | 12 months

SECONDARY OUTCOMES:
Number of patients alive at one-year post transplant | 12 months
Number of patients alive without recurrence of disease at one-year post transplant by conducting blood and bone marrow biopsy procedures | 12 months
Number of patients who died one year post-transplant not related to recurrence of disease | 12 months
Number of patients who fully engrafted (blood counts fully recovered) by conducting chimerism studies at 30-, 60-, 90-, 180-, and 365-days post transplant | 12 months
Number of patients who developed acute graft-versus-host disease by recording signs and symptoms of acute GVHD according to MAGIC standards at one-year post-transplant | 12 months
Number of patients who developed chronic graft-versus-host disease by recording signs and symptoms of chronic GVHD according to NIH standards at one-year post-transplant | 12 months
Number of patients who are alive at one-year post transplant who also did not develop GVHD | 12 months
Number of patients with treatment-related adverse events to venetoclax as assessed by CTCAE v5.0 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott Solomon, MD, Principal Investigator — Northside Hospital/BMTGA
Locations (1):
- Caitlin Guzowski, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Estey E, de Lima M, Tibes R, Pierce S, Kantarjian H, Champlin R, Giralt S. Prospective feasibility analysis of reduced-intensity conditioning (RIC) regimens for hematopoietic stem cell transplantation (HSCT) in elderly patients with acute myeloid leukemia (AML) and high-risk myelodysplastic syndrome (MDS). Blood. 2007 Feb 15;109(4):1395-400. doi: 10.1182/blood-2006-05-021907. Epub 2006 Oct 12. PMID 17038533
- [Result] Stelljes M, Beelen DW, Braess J, Sauerland MC, Heinecke A, Berning B, Kolb HJ, Holler E, Schwerdtfeger R, Arnold R, Spiekermann K, Muller-Tidow C, Serve HL, Silling G, Hiddemann W, Berdel WE, Buchner T, Kienast J; German AML Cooperative Group (AMLCG). Allogeneic transplantation as post-remission therapy for cytogenetically high-risk acute myeloid leukemia: landmark analysis from a single prospective multicenter trial. Haematologica. 2011 Jul;96(7):972-9. doi: 10.3324/haematol.2011.041004. Epub 2011 Apr 1. PMID 21459795
- [Result] Mawad R, Gooley TA, Sandhu V, Lionberger J, Scott B, Sandmaier BM, O'Donnell P, Becker PS, Petersdorf S, Dorcy KS, Hendrie P, Sorror ML, Walter RB, Deeg HJ, Appelbaum FR, Estey EH, Pagel JM. Frequency of allogeneic hematopoietic cell transplantation among patients with high- or intermediate-risk acute myeloid leukemia in first complete remission. J Clin Oncol. 2013 Nov 1;31(31):3883-8. doi: 10.1200/JCO.2013.50.2567. Epub 2013 Sep 23. PMID 24062388
- [Result] Medeiros BC, Satram-Hoang S, Hurst D, Hoang KQ, Momin F, Reyes C. Big data analysis of treatment patterns and outcomes among elderly acute myeloid leukemia patients in the United States. Ann Hematol. 2015 Jul;94(7):1127-38. doi: 10.1007/s00277-015-2351-x. Epub 2015 Mar 20. PMID 25791241
- [Result] Ostgard LSG, Lund JL, Norgaard JM, Norgaard M, Medeiros BC, Nielsen B, Nielsen OJ, Overgaard UM, Kallenbach M, Marcher CW, Riis AH, Sengelov H. Impact of Allogeneic Stem Cell Transplantation in First Complete Remission in Acute Myeloid Leukemia: A National Population-Based Cohort Study. Biol Blood Marrow Transplant. 2018 Feb;24(2):314-323. doi: 10.1016/j.bbmt.2017.10.019. Epub 2017 Oct 16. PMID 29051022
- [Result] Joshua TV, Rizzo JD, Zhang MJ, Hari PN, Kurian S, Pasquini M, Majhail NS, Lee SJ, Horowitz MM. Access to hematopoietic stem cell transplantation: effect of race and sex. Cancer. 2010 Jul 15;116(14):3469-76. doi: 10.1002/cncr.25297. PMID 20564154
- [Result] Landry I. Racial disparities in hematopoietic stem cell transplant: a systematic review of the literature. Stem Cell Investig. 2021 Dec 14;8:24. doi: 10.21037/sci-2021-058. eCollection 2021. PMID 35071585
- [Result] Abraham IE, Rauscher GH, Patel AA, Pearse WB, Rajakumar P, Burkart M, Aleem A, Dave A, Bharadwaj S, Paydary K, Acevedo-Mendez M, Goparaju K, Gomez R, Carlson K, Tsai SB, Quigley JG, Galvin JP, Zia M, Larson ML, Berg S, Stock W, Altman JK, Khan I. Structural racism is a mediator of disparities in acute myeloid leukemia outcomes. Blood. 2022 Apr 7;139(14):2212-2226. doi: 10.1182/blood.2021012830. PMID 35061876
- [Result] Bashey A, Zhang X, Morris LE, Holland HK, Bachier-Rodriguez L, Solomon SR, Solh M. Improved access to HCT with reduced racial disparities through integration with leukemia care and haploidentical donors. Blood Adv. 2023 Aug 8;7(15):3816-3823. doi: 10.1182/bloodadvances.2023009765. PMID 36961350
- [Result] Solomon SR, Sizemore CA, Zhang X, Brown S, Holland HK, Morris LE, Solh M, Bashey A. Impact of Donor Type on Outcome after Allogeneic Hematopoietic Cell Transplantation for Acute Leukemia. Biol Blood Marrow Transplant. 2016 Oct;22(10):1816-1822. doi: 10.1016/j.bbmt.2016.07.010. Epub 2016 Jul 21. PMID 27453362
- [Result] Fang M, Storer B, Estey E, Othus M, Zhang L, Sandmaier BM, Appelbaum FR. Outcome of patients with acute myeloid leukemia with monosomal karyotype who undergo hematopoietic cell transplantation. Blood. 2011 Aug 11;118(6):1490-4. doi: 10.1182/blood-2011-02-339721. Epub 2011 Jun 16. PMID 21680797
- [Result] Cornelissen JJ, Breems D, van Putten WL, Gratwohl AA, Passweg JR, Pabst T, Maertens J, Beverloo HB, van Marwijk Kooy M, Wijermans PW, Biemond BJ, Vellenga E, Verdonck LF, Ossenkoppele GJ, Lowenberg B. Comparative analysis of the value of allogeneic hematopoietic stem-cell transplantation in acute myeloid leukemia with monosomal karyotype versus other cytogenetic risk categories. J Clin Oncol. 2012 Jun 10;30(17):2140-6. doi: 10.1200/JCO.2011.39.6499. Epub 2012 May 7. PMID 22564995
- [Result] Middeke JM, Beelen D, Stadler M, Gohring G, Schlegelberger B, Baurmann H, Bug G, Bellos F, Mohr B, Buchholz S, Schwerdtfeger R, Martin H, Hegenbart U, Ehninger G, Bornhauser M, Schetelig J; Cooperative German Transplant Study Group. Outcome of high-risk acute myeloid leukemia after allogeneic hematopoietic cell transplantation: negative impact of abnl(17p) and -5/5q-. Blood. 2012 Sep 20;120(12):2521-8. doi: 10.1182/blood-2012-03-417972. Epub 2012 Jul 31. PMID 22855604
- [Result] Mohr B, Schetelig J, Schafer-Eckart K, Schmitz N, Hanel M, Rosler W, Frickhofen N, Link H, Neubauer A, Schuler U, Platzbecker U, Middeke JM, Ehninger G, Bornhauser M, Schaich M, Stolzel F; Study Alliance Leukaemia (SAL). Impact of allogeneic haematopoietic stem cell transplantation in patients with abnl(17p) acute myeloid leukaemia. Br J Haematol. 2013 Apr;161(2):237-44. doi: 10.1111/bjh.12253. Epub 2013 Feb 21. PMID 23432431
- [Result] Bowen D, Groves MJ, Burnett AK, Patel Y, Allen C, Green C, Gale RE, Hills R, Linch DC. TP53 gene mutation is frequent in patients with acute myeloid leukemia and complex karyotype, and is associated with very poor prognosis. Leukemia. 2009 Jan;23(1):203-6. doi: 10.1038/leu.2008.173. Epub 2008 Jul 3. No abstract available. PMID 18596741
- [Result] Seifert H, Mohr B, Thiede C, Oelschlagel U, Schakel U, Illmer T, Soucek S, Ehninger G, Schaich M; Study Alliance Leukemia (SAL). The prognostic impact of 17p (p53) deletion in 2272 adults with acute myeloid leukemia. Leukemia. 2009 Apr;23(4):656-63. doi: 10.1038/leu.2008.375. Epub 2009 Jan 8. PMID 19151774
- [Result] Lindsley RC, Saber W, Mar BG, Redd R, Wang T, Haagenson MD, Grauman PV, Hu ZH, Spellman SR, Lee SJ, Verneris MR, Hsu K, Fleischhauer K, Cutler C, Antin JH, Neuberg D, Ebert BL. Prognostic Mutations in Myelodysplastic Syndrome after Stem-Cell Transplantation. N Engl J Med. 2017 Feb 9;376(6):536-547. doi: 10.1056/NEJMoa1611604. PMID 28177873
- [Result] Poire X, Labopin M, Maertens J, Yakoub-Agha I, Blaise D, Ifrah N, Socie G, Gedde-Dhal T, Schaap N, Cornelissen JJ, Vigouroux S, Sanz J, Michaux L, Esteve J, Mohty M, Nagler A. Allogeneic stem cell transplantation in adult patients with acute myeloid leukaemia and 17p abnormalities in first complete remission: a study from the Acute Leukemia Working Party (ALWP) of the European Society for Blood and Marrow Transplantation (EBMT). J Hematol Oncol. 2017 Jan 18;10(1):20. doi: 10.1186/s13045-017-0393-3. PMID 28100265
- [Result] Loke J, Labopin M, Craddock C, Cornelissen JJ, Labussiere-Wallet H, Wagner-Drouet EM, Van Gorkom G, Schaap NPM, Kroger NM, Veelken JH, Rovira M, Menard AL, Bug G, Bazarbachi A, Giebel S, Brissot E, Nagler A, Esteve J, Mohty M. Additional cytogenetic features determine outcome in patients allografted for TP53 mutant acute myeloid leukemia. Cancer. 2022 Aug 1;128(15):2922-2931. doi: 10.1002/cncr.34268. Epub 2022 May 25. PMID 35612815
- [Result] Solomon SR, St Martin A, Shah NN, Fatobene G, Al Malki MM, Ballen KK, Bashey A, Bejanyan N, Bolanos Meade J, Brunstein CG, DeFilipp Z, Champlin RE, Fuchs EJ, Hamadani M, Hematti P, Kanakry CG, McGuirk JP, McNiece IK, Ciurea SO, Pasquini MC, Rocha V, Romee R, Patel SS, Vasu S, Waller EK, Wingard JR, Zhang MJ, Eapen M. Myeloablative vs reduced intensity T-cell-replete haploidentical transplantation for hematologic malignancy. Blood Adv. 2019 Oct 8;3(19):2836-2844. doi: 10.1182/bloodadvances.2019000627. PMID 31582392
- [Result] Solh MM, Solomon SR, Morris LE, Zhang X, Holland HK, Bashey A. The Dilemma of Conditioning Intensity: When Does Myeloablative Conditioning Improve Outcomes for Allogeneic Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2019 Mar;25(3):606-612. doi: 10.1016/j.bbmt.2018.09.012. Epub 2018 Sep 19. PMID 30244109
- [Result] Jin S, Cojocari D, Purkal JJ, Popovic R, Talaty NN, Xiao Y, Solomon LR, Boghaert ER, Leverson JD, Phillips DC. 5-Azacitidine Induces NOXA to Prime AML Cells for Venetoclax-Mediated Apoptosis. Clin Cancer Res. 2020 Jul 1;26(13):3371-3383. doi: 10.1158/1078-0432.CCR-19-1900. Epub 2020 Feb 13. PMID 32054729
- [Result] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- [Result] Valdez BC, Murray D, Yuan B, Nieto Y, Popat U, Andersson BS. ABT199/venetoclax potentiates the cytotoxicity of alkylating agents and fludarabine in acute myeloid leukemia cells. Oncotarget. 2022 Feb 10;13:319-330. doi: 10.18632/oncotarget.28193. eCollection 2022. PMID 35154579
- [Result] Garcia JS, Kim HT, Murdock HM, Cutler CS, Brock J, Gooptu M, Ho VT, Koreth J, Nikiforow S, Romee R, Shapiro R, Loschi F, Ryan J, Fell G, Karp HQ, Lucas F, Kim AS, Potter D, Mashaka T, Stone RM, DeAngelo DJ, Letai A, Lindsley RC, Soiffer RJ, Antin JH. Adding venetoclax to fludarabine/busulfan RIC transplant for high-risk MDS and AML is feasible, safe, and active. Blood Adv. 2021 Dec 28;5(24):5536-5545. doi: 10.1182/bloodadvances.2021005566. PMID 34614506
- [Result] Valdez BC, Tang X, Li Y, Murray D, Liu Y, Popat U, Champlin RE, Andersson BS. Epigenetic modification enhances the cytotoxicity of busulfan and4-hydroperoxycyclophosphamide in AML cells. Exp Hematol. 2018 Nov;67:49-59.e1. doi: 10.1016/j.exphem.2018.08.002. Epub 2018 Aug 10. PMID 30102945